CLINICAL TRIAL: NCT03169127
Title: Clinical Pharmacogenetic of Ibuprofen Enantiomers After Lower Third Molar Surgeries
Brief Title: Clinical Pharmacogenetic of Ibuprofen After Lower Third Molar Surgeries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Giovana Maria Weckwerth, DDS, PhD student, Principal Investigator, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 59807716.9.0000.5417
Record Dates: First submitted 2017-03-16; First posted 2017-05-30 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Pain; Other Surgical Procedures; Impacted Third Molar Tooth
Keywords: Ibuprofen; Lower third molar; Oral Surgery
MeSH Terms: conditions — Pain | interventions — Ibuprofen; Pharmacogenomic Testing

STUDY DESIGN:
Intervention Model Description: Two Hundred healthy volunteers underwent removal of one lower third molar, will be treated to control pain, swelling and trismus with ibuprofen 600mg. Therefore, these 200 patients will be genotyped and phenotyped for these genes and their postoperative records with all data collected will be compared with the haplotypes found in the Brazilian population.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Group Ibuprofen 600mg (Experimental): Two Hundred healthy volunteers underwent removal of one lower third molar, will be treated to control pain, swelling and trismus with ibuprofen 600mg. Therefore, these 200 patients will be genotyped and phenotyped for these genes and their postoperative records with all data collected will be compared with the haplotypes found in the Brazilian population.
  Interventions: Drug: Ibuprofen 600 mg

INTERVENTIONS:
Drug: Ibuprofen 600 mg — After lower third molars surgeries, pharmacogenetic and clinical efficacy of Ibuprofen 600mg was study.
  Other Names: Lower third molar surgery with ibuprofen for pharmacogenetic

SUMMARY:
The present clinical trial randomized will be to assess the link between the different haplotypes of CYP2C8 and CYP2C9 genes and the clinical efficacy of ibuprofen after lower third molar extractions. Onset, duration of postoperative analgesia, duration of anesthetic action on soft tissues, intraoperative bleeding, hemodynamic parameters, postoperative mouth opening and wound healing at the 7th postoperative day were evaluated. For this purpose, 200 healthy volunteers underwent removal of one lower third molar, under local anesthesia with articaine 4% (1:200,000 adrenaline) will be genotyped and phenotyped for these genes and their postoperative records with all data collected will be compared with the haplotypes found in the Brazilian population.

DETAILED DESCRIPTION:
The aim of this study will be to assess the link between the different haplotypes of CYP2C8 and CYP2C9 genes and the clinical efficacy of ibuprofen after lower third molar extractions regarding pain, swelling and trismus, adverse reactions, the amount of pain medication used, the patient satisfaction with the drug and the influence of the ability on preoperative modulation of conditioned pain. We will evaluate also the relationship between the different haplotypes of OPRM1 gene (SNP A118G), the salivary concentrations of pro-inflammatory cytokines (IL-2, IL-4, IL-6, IL-10 and TNF-±), and preoperative conditioned pain modulation. Therefore, 200 patients will be genotyped and phenotyped for these genes and their postoperative records with all data collected will be compared with the haplotypes found in the Brazilian population.

For analysis of the proposed genes, saliva will be collected, which will serve as a source of genomic DNA. For molecular analysis it will be performed polymerase chain reaction (PCR). All tests will be conducted and validated by Applied Biosystems®. Also it will be held in the research, genetic sequencing of the genes CYP2C8, CYP2C9 and OPRM1, to verify possible correlations of these genes with postoperative pain and pain modulation.

ELIGIBILITY:
Inclusion Criteria:

* Need of lower third molar surgeries

Exclusion Criteria:

* Presence of systemic diseases;
* Presence of local inflammation and/or infection;
* Any history of allergic reaction to local anesthetics, gastrointestinal bleeding or ulceration;
* Cardiovascular, kidney or hepatic diseases;
* Patients who are making use of antidepressants, diuretics or anticoagulants;
* Asthma and allergy to aspirin, ibuprofen or any other nonsteroidal antiinflammatory drug;
* Regular use of any nonsteroidal antiinflammatory drug,
* Pregnancy or breast feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of changes in the postsurgical pain during the first 24 hours until 96 hours after the procedure | Seventh postoperative day
  Subjective evaluation of postsurgical pain, which was annotated by the volunteer after the surgery, in a Visual Analogue Scale (VAS, 0-100 mm). The subjective pain evaluations will be performed by patients at the following times after administration of the drug [0, 15, 30 and 45 min, 1; 1.5; 2; 3; 4; 5; 6; 7; 8; 10; 12; 16; 24 hr, 48, 72 and 96 h]. What will be taken into account on this outcome is the representation of the postsurgical pain, that will be noted on the Visual Analogue Scale (in millimeters) in respective moments.
Quality of anesthesia | During the surgical procedure
  Quality of anesthesia during surgery based on a category 3point scale: 1) the patient reported no discomfort; 2) the patient reported discomfort, without the need to supplement the anesthesia; 3) reported some discomfort by the patient, requiring anesthesia complementation. Intraoral bleeding that will be evaluated by the surgeon according to a 3point scale (1: minimal, 2: normal and 3: Maximum), immediately after the following steps: injection of the first cartridge anesthesia, incision, mucoperiosteal detachment, osteotomies, tooth section, extraction, cleaning and suturing.
Intraoperative bleeding during the surgeries steps | During the surgical procedure
  Intraoperative bleeding, rated by the surgeon according to a 3 point category rating scale (1 minimal bleeding; 2 normal bleeding; 3 excessive bleeding) (SISK, 1986), immediately after the following steps: injection of the first cartridge of articaine, tissue incision, flap reflection, bone removal (when this procedure was necessary), tooth extraction, cleaning of the operated site, and completion of suturing.
Blood pressure variability during the surgeries steps | During the surgical procedure
  Systolic blood pressure, diastolic, and mean to be verified and recorded at surgical moments previously described (injection of the first cartridge anesthesia, incision, mucoperiosteal detachment, osteotomies, tooth section, extraction, cleaning and suturing), carried out with the aid of a system for monitoring hemodynamic parameters.
Heart rate variability during the surgeries steps | During the surgical procedure
  Heart rate to be verified and recorded surgical at moments described above, carried out with the aid of a system for monitoring hemodynamic parameters.
Oxygen saturation variability during the surgeries steps | During the surgical procedure
  Oxygen saturation to be verified and recorded at surgical moments described above, carried out with the aid of a system for monitoring hemodynamic parameters.
Subjective evaluation of postsurgical pain at the moment of the rescue medication utilization | Seventh postoperative day
  Subjective evaluation of postsurgical pain at the moment of the rescue medication consumption which was annotated by the volunteer after the surgery, in a Visual Analogue Scale (VAS, 0-100 mm).

SECONDARY OUTCOMES:
Postoperative mouth opening | Second and Seventh postoperative days
  Mouth opening (mm) between the mesial-incisal corners of the upper and lower right central incisors at maximum opening of the jaws was measured and recorded before the surgery and during the second and seventh postoperative days.
Onset and duration of surgery after administration of local anesthetic | During the surgery
  Will only be considered those surgeries in which there is no difference in the duration time of the procedure between the patients. This time count will be started after the administration of the first local anesthetic. Unit of mesure used will be hours.
Incidence, type and severity of adverse reactions after the surgery | Seventh postoperative day
  Will be considered as adverse reactions: gastrointestinal irritation, nausea, vomiting, bleeding, allergy, headache, dizziness, drowsiness or any other type of reaction presented after surgery.
Total amount of rescue medication | Seventh postoperative day
  The total amount of rescue medication that was used by the patient during the postoperative period (Acetominophen- 750 mg) will be analyzed.
Measurement the facial edema | On the second day after surgery and on the seventh day after surgery.
  It will apply the method used by Ustun et al. (2003), which takes into account the sum of the following measures (obtained with flexible tape measure): A) distance between the lateral corner of the eye and the gonion, B) away from the tragus corner of the mouth and C) away from the tragus to the soft tissue of pogonion. Preoperative sum of three measures will be considered as the baseline that way. The difference between the values obtained in the postoperative period and baseline indicate the facial edema in the 2nd and 7th days.

CONTACTS AND LOCATIONS:
Overall Officials: Giovana M Weckwerth, DDS, Principal Investigator — 416.016.638-54
Locations (1):
- University of São Paulo, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weckwerth GM, Dionisio TJ, Costa YM, Zupelari-Goncalves P, Oliveira GM, Torres EA, Bonjardim LR, Faria FAC, Calvo AM, Moore T, Absher DM, Santos CF. Multifocal Analysis of Acute Pain After Third Molar Removal. Front Pharmacol. 2021 Apr 15;12:643874. doi: 10.3389/fphar.2021.643874. eCollection 2021. PMID 33935738
- [Derived] Weckwerth GM, Dionisio TJ, Costa YM, Colombini-Ishiquiriama BL, Oliveira GM, Torres EA, Bonjardim LR, Calvo AM, Moore T, Absher DM, Santos CF. CYP450 polymorphisms and clinical pharmacogenetics of ibuprofen after lower third molar extraction. Eur J Clin Pharmacol. 2021 May;77(5):697-707. doi: 10.1007/s00228-020-03046-0. Epub 2020 Nov 17. PMID 33205280